CLINICAL TRIAL: NCT00765882
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Trial of Linaclotide Administered Orally for 12 Weeks in Patients With Chronic Constipation
Brief Title: Phase III, Randomized, Double-Blind, Placebo-Controlled, Trial of Linaclotide Administered to Patients With Chronic Constipation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Collaborators: Ironwood Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LIN-MD-01
Record Dates: First submitted 2008-10-01; First posted 2008-10-03 (Estimated); Results first posted 2013-01-30 (Estimated); Last update posted 2013-01-30 (Estimated); Status verified 2012-12

CONDITIONS: Chronic Constipation
Keywords: Constipation; Chronic Constipation; Linaclotide
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- 1 (Experimental): Linaclotide 290 micrograms
  Interventions: Drug: Linaclotide 290 micrograms
- 2 (Experimental): Linaclotide 145 micrograms
  Interventions: Drug: Linaclotide 145 micrograms
- 3 (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Linaclotide 290 micrograms — Oral, once daily each morning at least 30 minutes before breakfast for the duration of the study
  Arms: 1
Drug: Linaclotide 145 micrograms — Oral, once daily each morning at least 30 minutes before breakfast for the duration of the study
  Arms: 2
Drug: Placebo — Oral, once daily each morning at least 30 minutes before breakfast for the duration of the study
  Arms: 3

SUMMARY:
The objective of this trial is to determine the efficacy and safety of linaclotide administered to patients with chronic constipation (CC). The primary efficacy parameter is the percentage of patients in each treatment group that meet the protocol definition for Complete Spontaneous Bowel Movement (CSBM) Overall Responder

ELIGIBILITY:
Inclusion Criteria:

* Patient has completed a colonoscopy according to the AGA criteria, with no clinically significant findings
* Patient has successfully completed protocol procedures (with no clinically significant findings): physical exam, 12-lead ECG, or clinical laboratory tests
* Patient meets protocol criteria for CC: reports < 3 bowel movements per week and reports straining, lumpy or hard stools, and/or sensation of incomplete evacuation during > 25% of BMs
* Patient demonstrates continued chronic constipation through Pretreatment Period
* Patient is compliant with IVRS

Exclusion Criteria:

* Patient has history of loose or watery stools
* Patient has symptoms of or been diagnosed with Irritable Bowel Syndrome (IBS)
* Patient has a structural abnormality of the gastrointestinal (GI) tract or a disease or condition that can affect GI motility
* Patient has any protocol-excluded or clinically significant medical or surgical history that could confound the study assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 633 (Actual)
Dates: Start 2008-09; Primary Completion 2009-07 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul F.C. Eng, PhD, Study Director — Forest Laboratories
Locations (100):
- United States (92):
  - Forest Investigative Site, Birmingham, Alabama
  - Forest Investigative Site, Huntsville, Alabama
  - Forest Investigative Site, Chandler, Arizona
  - Forest Investigative Site, Mesa, Arizona
  - Forest Investigative Site, Peoria, Arizona
  - Forest Investigative Site, Phoenix, Arizona
  - Forest Investigative Site, Scottsdale, Arizona
  - Forest Investigative Site, Tucson, Arizona
  - Forest Investigative Site, Burbank, California
  - Forest Investigative Site, Encinitas, California
  - Forest Investigative Site, Foothill Ranch, California
  - Forest Investigative Site, Los Angeles, California
  - Forest Investigative Site, Orange, California
  - Forest Investigative Site, Westlake Village, California
  - Forest Investigative Site, Boulder, Colorado
  - Forest Investigative Site, Colorado Springs, Colorado
  - Forest Investigative Sites, Denver, Colorado
  - Forest Investigative Site, Longmont, Colorado
  - Forest Investigative Site, Wheat Ridge, Colorado
  - Forest Investigative Site, Waterbury, Connecticut
  - Forest Investigative Site, Boca Raton, Florida
  - Forest Investigative Site, Bradenton, Florida
  - Forest Investigative Site, Brooksville, Florida
  - Forest Investigative Site, Fort Myers, Florida
  - Forest Investigative Site, Jupiter, Florida
  - Forest Investigative Site, Kissimmee, Florida
  - Forest Investigative Site, Miami, Florida
  - Forest Investigative Site, Ocala, Florida
  - Forest Investigative Site, Orlando, Florida
  - Forest Investigative Site, Panama City, Florida
  - Forest Investigative Site, Pembroke Pines, Florida
  - Forest Investigative Site, St. Petersburg, Florida
  - Forest Investigative Site, Tampa, Florida
  - Forest Investigative Site, Trinity, Florida
  - Forest Investigative Site, Zephyrhills, Florida
  - Forest Investigative Site, Atlanta, Georgia
  - Forest Investigative Site, Marietta, Georgia
  - Forest Investigative Site, Stockbridge, Georgia
  - Forest Investigative Site, Woodstock, Georgia
  - Forest Investigative Site, Idaho Falls, Idaho
  - Forest Investigative Site, Rockford, Illinois
  - Forest Investigative Site, Elkhart, Indiana
  - Forest Investigative Site, Evansville, Indiana
  - Forest Investigative Site, Indianapolis, Indiana
  - Forest Investigative Site, Iowa City, Iowa
  - Forest Investigative Site, Arkansas City, Kansas
  - Forest Investigative Site, Newton, Kansas
  - Forest Investigative Site, Wichita, Kansas
  - Forest Investigative Site, Lexington, Kentucky
  - Forest Investigative Site, Madisonville, Kentucky
  - Forest Investigative Site, Chevy Chase, Maryland
  - Forest Investigative Site, Hagerstown, Maryland
  - Forest Investigative Site, Lutherville, Maryland
  - Forest Investigative Site, Boston, Massachusetts
  - Forest Investigative Site, Chaska, Minnesota
  - Forest Investigative Site, St Louis, Missouri
  - Forest Investigative Site, Vineland, New Jersey
  - Forest Investigative Site, Albuquerque, New Mexico
  - Forest Investigative Site, Brooklyn, New York
  - Forest Investigative Site, Great Neck, New York
  - Forest Investigative Site, Fayetteville, North Carolina
  - Forest Investigative Site, Greensboro, North Carolina
  - Forest Investigative Site, Hickory, North Carolina
  - Forest Investigative Site, Raleigh, North Carolina
  - Forest Investigative Site, Wilmington, North Carolina
  - Forest Investigative Site, Winston-Salem, North Carolina
  - Forest Investigative Site, Bismarck, North Dakota
  - Forest Investigative Site, Akron, Ohio
  - Forest Investigative Site, Cincinnati, Ohio
  - Forest Investigative Site, Cleveland, Ohio
  - Forest Investigative Site, Oklahoma City, Oklahoma
  - Forest Investigative Site, Tulsa, Oklahoma
  - Forest Investigative Site, Bensalem, Pennsylvania
  - Forest Investigative Site, Pittsburgh, Pennsylvania
  - Forest Investigative Site, Greenville, South Carolina
  - Forest Investigative Site, Greer, South Carolina
  - Forest Investigative Site, Nashville, Tennessee
  - Forest Investigative Site, Austin, Texas
  - Forest Investigative Site, Dallas, Texas
  - Forest Investigative Site, Houston, Texas
  - Forest Investigative Site, Lake Jackson, Texas
  - Forest Investigative Site, San Antonio, Texas
  - Forest Investigative Site, Salt Lake City, Utah
  - Forest Investigative Site, Charlottesville, Virginia
  - Forest Investigative Site, Christianburg, Virginia
  - Forest Investigative Site, Newport News, Virginia
  - Forest Investigative Site, Norfolk, Virginia
  - Forest Investigative Site, Richmond, Virginia
  - Forest Investigative Site, Bellevue, Washington
  - Forest Investigative Site, Lakewood, Washington
  - Forest Investigative Site, Wenatchee, Washington
  - Forest Investigative Site, Milwaukee, Wisconsin
- Canada (8):
  - Forest Investigative Site, Vancouver, British Columbia
  - Forest Investigative Site, Greater Sudbury, Ontario
  - Forest Investigative Site, Hamilton, Ontario
  - Forest Investigative Site, Newmarket, Ontario
  - Forest Investigative Site, Ottawa, Ontario
  - Forest Investigative Site 1, Sarnia, Ontario
  - Forest Investigative Site 2, Sarnia, Ontario
  - Forest Investigative Site, Toronto, Ontario

REFERENCES:
- [Derived] Chang L, Lembo AJ, Lavins BJ, Shiff SJ, Hao X, Chickering JG, Jia XD, Currie MG, Kurtz CB, Johnston JM. The impact of abdominal pain on global measures in patients with chronic idiopathic constipation, before and after treatment with linaclotide: a pooled analysis of two randomised, double-blind, placebo-controlled, phase 3 trials. Aliment Pharmacol Ther. 2014 Dec;40(11-12):1302-12. doi: 10.1111/apt.12985. Epub 2014 Oct 13. PMID 25312449
- [Derived] Lembo AJ, Schneier HA, Shiff SJ, Kurtz CB, MacDougall JE, Jia XD, Shao JZ, Lavins BJ, Currie MG, Fitch DA, Jeglinski BI, Eng P, Fox SM, Johnston JM. Two randomized trials of linaclotide for chronic constipation. N Engl J Med. 2011 Aug 11;365(6):527-36. doi: 10.1056/NEJMoa1010863. PMID 21830967

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient Recruitment occurred from October 2008 to March 2009 at 103 study centers (95 in the United States and 8 in Canada).
Pre-assignment Details: Patients went through a 14 to 21 day Pretreatment Period during which the patients provided qualifying bowel habit and symptoms, and rescue medicine usage information through an interactive voice response system (IVRS).
Groups:
- Placebo: Dose matched placebo, oral administration, once per day.
- Linaclotide 145µg: Linaclotide, 145µg dose, oral administration, once per day
- Linaclotide 290µg: Linaclotide, 290µg dose, oral administration, once per day
Period: Overall Study
Arm/Group | Placebo | Linaclotide 145µg | Linaclotide 290µg
Started | 215 | 213 | 205
Completed | 191 | 173 | 169
Not Completed | 24 | 40 | 36
Not completed — Adverse Event | 10 | 21 | 20
Not completed — Lack of Efficacy | 4 | 0 | 1
Not completed — Protocol Violation | 4 | 3 | 1
Not completed — Withdrawal by Subject | 2 | 6 | 6
Not completed — Lost to Follow-up | 1 | 9 | 6
Not completed — Other Reason | 3 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Linaclotide 145µg | Linaclotide 290µg | Total
Number analyzed (Participants) | 215 | 213 | 205 | 633
Age Continuous [Mean (Standard Deviation); unit: years] | 47.0 (13.5) | 48.5 (12.3) | 47.3 (13.3) | 47.6 (13.0)
Age, Customized [Number; unit: participants]
  18 years to 64 years | 188 | 189 | 183 | 560
  65 years and older | 27 | 24 | 22 | 73
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 196 | 195 | 181 | 572
  Male | 19 | 18 | 24 | 61
Region of Enrollment [Number; unit: participants]
  United States | 208 | 208 | 198 | 614
  Canada | 7 | 5 | 7 | 19

OUTCOME MEASURES:

1. Primary Outcome: Complete Spontaneous Bowel Movement (CSBM) Overall Responder
Description: A 12-week CSBM overall responders was defined as a patient who for at least 9 of the 12 weeks of the treatment period had a CSBM weekly frequency rate that was 3 or greater and increased by 1 or more from baseline.
  A CSBM was defined as a spontaneous bowel movement (SBM) that was associated with a sense of complete evacuation.
  An SBM was defined as a bowel movement (BM) that occurred in the absence of laxative, enema, or suppository use on either the calendar day of the BM or the calendar day before the BM.
Time Frame: Change from Baseline to Week 12
Population: A total of 633 patients were randomized to treatment and received at least 1 dose of study drug. 630 patients were included in the Intent to Treat (ITT) Population. An observed-cases approach to missing postbaseline data was applied.
Measure: Number; unit: participants
Arm/Group | Placebo | Linaclotide 145µg | Linaclotide 290µg
Number analyzed (Participants) | 215 | 213 | 202
participants
  Responder | 13 | 34 | 43
  Nonresponder | 202 | 179 | 159
Statistical Analysis 1: Comparison: Placebo vs Linaclotide 145µg; Null hypothesis: There is no difference in the proportion of 12-week CSBM overall responders between patients taking the 145-μg dose and those taking placebo. The power, adjusted for multiplicity, was expected to be 90% based on study NCT00402337 (MCP-103-201) data; Test type: Superiority or Other; p = 0.0012, Cochran-Mantel-Haenszel — The p-value is still less than 0.05 after adjusting multiplicity using a serial gatekeeping multiple comparison procedure; Odds Ratio (OR) = 2.93, 95% CI 2-sided [1.50 to 5.72]
Statistical Analysis 2: Comparison: Placebo vs Linaclotide 290µg; Null hypothesis: There is no difference in the proportion of 12-week CSBM overall responders between patients taking the 290-μg dose and those taking placebo. The power, adjusted for multiplicity, was expected to be 96% based on study NCT00460811 (MCP-103-202) data; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 4.22, 95% CI 2-sided [2.20 to 8.10]

2. Secondary Outcome: 12-week Complete Spontaneous Bowel Movement (CSBM) Frequency Rate
Description: The number of CSBMs per week.
Time Frame: Change from Baseline to Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: CSBM per week
Arm/Group | Placebo | Linaclotide 145µg | Linaclotide 290µg
Number analyzed (Participants) | 215 | 213 | 202
CSBM per week | 0.614 (0.209) | 2.011 (0.215) | 2.653 (0.217)

3. Secondary Outcome: 12-Week Spontaneous Bowel Movement (SBM) Frequency Rate
Description: A patient's 12-week spontaneous bowel movement (SBM) frequency rate was the number of SBMs per week calculated over the 12-weeks of the treatment period.
Time Frame: Change from Baseline to Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: SBM per week
Arm/Group | Placebo | Linaclotide 145µg | Linaclotide 290µg
Number analyzed (Participants) | 215 | 213 | 202
SBM per week | 1.113 (0.265) | 3.466 (0.272) | 3.675 (0.275)

4. Secondary Outcome: 12-Week Stool Consistency
Description: The consistency of each BM was assessed using the 7-point Bristol Stool Form Scale:
  1. = separate hard lumps like nuts [difficult to pass]
  2. = sausage shaped but lumpy
  3. = like a sausage but with cracks on surface
  4. = like a sausage or snake, smooth and soft
  5. = soft blobs with clear-cut edges [passed easily]
  6. = fluffy pieces with ragged edges, a mushy stool
  7. = watery, no solid pieces [entirely liquid]
Time Frame: Change from Baseline to Week 12
Population: A total of 633 patients were randomized to treatment and received at least 1 dose of study drug. 630 patients were included in the ITT Population; 97 patients with no pretreatment spontaneous bowel movements were excluded from the 12-Week Stool Consistency analysis. An observed-cases approach to missing postbaseline data was applied.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Linaclotide 145µg | Linaclotide 290µg
Number analyzed (Participants) | 183 | 182 | 168
units on a scale | 0.572 (0.098) | 1.823 (0.100) | 2.009 (0.103)

5. Secondary Outcome: 12-Week Severity of Straining
Description: Straining is measured on a 5-point scale, where a value of 1 is "not at all" and a value of 5 is "an extreme amount.
Time Frame: Change from Baseline to Week 12
Population: A total of 633 patients were randomized to treatment and received at least 1 dose of study drug. 630 patients were included in the ITT Population; 97 Patients with no pretreatment spontaneous bowel movements were excluded from the 12-Week Severity of Straining analysis. An observed-cases approach to missing postbaseline data was applied.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Linaclotide 145µg | Linaclotide 290µg
Number analyzed (Participants) | 183 | 182 | 168
units on a scale | -0.554 (0.060) | -1.141 (0.061) | -1.208 (0.063)

6. Secondary Outcome: 12-Week Abdominal Discomfort
Description: Abdominal discomfort is based on a 5-point scale where a value of l is "none" and a value of 5 is "very severe."
Time Frame: Change from Baseline to Week 12
Population: A total of 633 patients were randomized to treatment and received at least 1 dose of study drug. 630 patients were included in the Intent to Treat (ITT) Population. 1 additional patient without a baseline Abdominal Discomfort score was excluded from analysis in this endpoint. An observed-cases approach to missing postbaseline data was applied.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Linaclotide 145µg | Linaclotide 290µg
Number analyzed (Participants) | 215 | 213 | 201
units on a scale | -0.271 (0.043) | -0.455 (0.044) | -0.485 (0.045)

7. Secondary Outcome: 12-Week Bloating
Description: Bloating was based on a 5-point scale where a value of l is "none" and a value of 5 is "very severe".
Time Frame: Change from Baseline to Week 12
Population: A total of 633 patients were randomized to treatment and received at least 1 dose of study drug. 630 patients were included in the ITT population; 1 additional patient without a baseline Bloating score was excluded from analysis in this endpoint. An observed-cases approach to missing postbaseline data was applied.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Linaclotide 145µg | Linaclotide 290µg
Number analyzed (Participants) | 215 | 213 | 201
units on a scale | -0.244 (0.048) | -0.432 (0.049) | -0.485 (0.049)

8. Secondary Outcome: 12-Week Constipation Severity
Description: Constipation severity was based on a 5-point ordinal scale where a value of l is "none" and a value of 5 is "very severe".
Time Frame: Change from Baseline to Week 12
Population: A total of 633 patients were randomized to treatment and received at least 1 dose of study drug. 630 patients were included in the ITT population; 11 additional patients who dropped out prior to finishing 1 week of the trial were excluded from the Constipation Severity endpoint. An observed-cases approach to missing postbaseline data was applied.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Linaclotide 145µg | Linaclotide 290µg
Number analyzed (Participants) | 212 | 209 | 198
units on a scale | -0.306 (0.062) | -0.908 (0.063) | -0.954 (0.064)

ADVERSE EVENTS:
Time Frame: Adverse Event reporting occurred from October 2008 through August 2009.
Arm/Group | Placebo | Linaclotide 145µg | Linaclotide 290µg
Serious Adverse Events (participants affected / at risk) | 4/215 | 3/213 | 7/205
Other Adverse Events (participants affected / at risk) | 35/215 | 70/213 | 49/205
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=215) | Linaclotide 145µg (N=213) | Linaclotide 290µg (N=205)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Diverticulitis (Gastrointestinal disorders) | 0 | 0 | 1
Drug toxicity (Injury, poisoning and procedural complications) | 0 | 1 | 0
Endometriosis (Reproductive system and breast disorders) | 0 | 0 | 1
Lymphoma (Blood and lymphatic system disorders) | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Postoperative wound infection (Injury, poisoning and procedural complications) | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0
Cellulitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Goitre (Endocrine disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=215) | Linaclotide 145µg (N=213) | Linaclotide 290µg (N=205)
Diarrhea (Gastrointestinal disorders) | 6 | 42 | 30
Flatulence (Gastrointestinal disorders) | 13 | 16 | 13
Upper respiratory tract infection (Infections and infestations) | 14 | 16 | 9
Abdominal pain (Gastrointestinal disorders) | 5 | 11 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data generated in this study will be the property of Forest Research Institute. An integrated clinical and statistical report will be prepared at the completion of the trial. Publication of the results by the Investigator will be subject to mutual agreement between the Investigator and Forest Research Institute